CLINICAL TRIAL: NCT05356000
Title: Determine the Contribution of Paracellular GI Oxalate Absorption in Obese and Roux-en-Y Gastric Bypass Kidney Stone Patients
Brief Title: GI Oxalate Absorption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB22-0023
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Bariatric Surgery Candidate; Kidney Stone
Keywords: Roux-en-Y Gastric Bypass; RYGB; Oxalate
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects who will follow low-oxalate diet followed by visit to research clinic (Other): 30 stone-forming participants will be recruited to this study.
  Interventions: Other: Special low-oxalate diet followed by all-day visit to University of Chicago research clinic

INTERVENTIONS:
Other: Special low-oxalate diet followed by all-day visit to University of Chicago research clinic — Active participation in this study will last for around one week. For the first two days, participants will be asked to eat a special diet at home. From Days 3-5, they will eat special meals that will be delivered to their home from a research clinic at the University of Chicago. They will also collect urine at home on Days 4 and 5.
  On Day 6, subjects will come in to the research clinic at the University of Chicago in Hyde Park, where they will spend most of the day. They will receive a special liquid that contains oxalate, and will receive a specially prepared breakfast that is low in oxalate and citrate. After this, we will collect their urine and blood throughout the day. We will draw blood 4 separate times.

SUMMARY:
This study aims to learn more about how oxalate, a compound found in many foods, may affect a person's chances of forming kidney stones. Active participation in this study will last for around one week.

For the first two days, subjects will be asked to eat a special diet at home. From Days 3-5, they will eat special meals delivered to their home from a research clinic at the University of Chicago. They will also collect 24-hour urine samples at home on Days 4 and 5. On Day 6, they will come in to the research clinic at the University of Chicago in Hyde Park, where they will spend most of the day. They will receive a special liquid that contains oxalate, and we will have them eat a specially prepared breakfast that is low in oxalate and citrate.

DETAILED DESCRIPTION:
The study will be carried out in the University of Chicago Medicine (UCM) Clinical Research Center (CRC).

Study Population and Recruitment Enroll 10 post-Roux-en-Y Gastric Bypass stone forming, 10 obese stone forming, and 10 non-obese stone forming participants over four years of the award. Patients will be recruited at the University of Chicago Kidney Stone Clinic and Bariatric Surgery Clinics (both current and repository of previous patients). The Bariatric Surgery Clinic is a large clinic and Center for Excellence for bariatric surgery. The group's four active surgeons (including study advisor, Dr. John Alverdy) perform 300 bariatric surgeries per year. Over the past 10 years, at least one quarter to one half of these procedures have been Roux-en-Y Gastric Bypass. Incidence rates for stones at 10 years after Roux-en-Y Gastric Bypass is 14% and thus, even with conservative estimates, we will have over 100 eligible patients from this clinic.

Experimental Design and Implications Administration of very low oxalate diet (50mg/day) for three days followed by 13c2-oxalate and sucralose oral load test will determine the amount of oxalate absorbed via gastrointestinal (GI) paracellular pathways discriminated from endogenous oxalate production. Urine oxalate levels after low oxalate diet will provide an estimate of GI oxalate absorption combined with hepatic production (Aim 2a). By measuring the proportion of 13c2-oxalate load that appears in the urine, we will determine the fraction of absorbed oxalate that appears in the urine. Sucralose will be used with the load test as a marker of paracellular transport. Sucralose is an artificial sweetener that is absorbed in the GI tract via paracellular pathways and excreted unchanged in the urine. It is used to estimate permeability of the whole GI tract and as a marker of paracellular GI transport. Along with 13c2-oxalate, sucralose has been used to study GI oxalate transport mechanisms.

The knowledge obtained from these studies will determine the contribution of GI absorption of dietary oxalate and how it is absorbed from the GI tract. These data will provide crucial information to understanding mechanisms for stone risk in obese and Roux-en-Y Gastric Bypass stone formers. If high urine oxalate in Roux-en-Y Gastric Bypass and obese stone forming is primarily due to GI hyperabsorption, then a low oxalate diet will not decrease urine oxalate levels and levels will decrease less in obese and Roux-en-Y Gastric Bypass stone formers than non-obese stone formers. This will potentially reset the clinical utility of a low oxalate diet in these patients. If high urine oxalate is from GI paracellular hyperabsorption, then the percent absorption of 13c2-oxalate and sucralose will be greater in obese and post-Roux-en-Y Gastric Bypass stone formers compared with non-obese stone formers. Follow up studies will focus on how to block or blunt this mechanism. If high urine oxalate in obese and Roux-en-Y Gastric Bypass stone forming is due to other oxalate sources (i.e. endogenous production) then the percent absorption of 13c2-oxalate and sucralose will not be greater in obese and Roux-en-Y Gastric Bypass stone formers compared with non-obese stone formers. Clinically, this will direct patients and physicians towards higher impact management strategies with less emphasis on a low oxalate diet. Future studies will investigate endogenous production of oxalate in obese and Roux-en-Y Gastric Bypass stone formers. Better strategies for oxalate management after surgery will lower kidney stone risk in these high-risk patients and lower the risk of chronic kidney disease progression and end-stage renal disease that can result from high urine oxalate.

In non-obese stone formers (N=10) obese stone formers (N=10) and post-Roux-en-Y Gastric Bypass stone formers (N=10), we will measure urine oxalate and citrate before and after three days of low (50mg/day) oxalate diet. Primary endpoint (hypothesis 2a) is change in urine oxalate excretion from baseline after low oxalate diet in non-obese versus obese and Roux-en-Y Gastric Bypass stone formers. 2b and 2c: Following the low oxalate diet, give a 13c2-labeled sodium oxalate (100mg) and sucralose (5g) oral load test and measure urine oxalate, citrate, and sucralose over 24 hours. Primary endpoint (hypothesis 2b) is percent 13c2-oxalate of total administered in non-obese versus obese and Roux-en-Y Gastric Bypass stone formers. Secondary endpoint (hypothesis 2c) is percent sucralose of total administered in non-obese versus obese and Roux-en-Y Gastric Bypass stone formers.

Rationale: Absorption of diet oxalate may be elevated in obese and post-Roux-en-Y Gastric Bypass stone formers, however the actual contribution of increased gastrointestinal (GI) oxalate absorption to hyperoxaluria in these patients has not been documented. It is also unclear what proportion of oxalate is absorbed via the paracellular route. If an increase in GI oxalate absorption is not sufficient to explain hyperoxaluria, it would change treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

Post-Roux-en-Y gastric bypass stone formers:

* Age 18-70
* Previous history of Roux-en-Y gastric bypass
* History of at least one calcium-based kidney stone after surgery
* Pre-protocol urine oxalate above the lab normal range (50mg/day)

Obese stone formers:

* Age 18-70
* Body mass index (BMI) >=30kg/m2
* History of at least one calcium-based kidney stone
* Pre-protocol urine oxalate above the lab normal range (50mg/day)

Non-obese stone formers:

* Age 18-70, BMI between 18.5-29.9 kg/m2
* History of at least one calcium-based kidney stone

Exclusion Criteria:

Post-Roux-en-Y gastric bypass stone formers:

* History of colon resection (partial or complete)
* History of duodenal switch bowel surgery
* History of ileal-jejunal bypass surgery
* History of primarily uric acid, cysteine, or struvite stones

Obese and non-obese stone formers:

* History of bowel surgery
* History of colon resection
* History of inflammatory bowel disease (Crohn's disease, Ulcerative Colitis)
* History of primarily uric acid, cysteine, or struvite stones

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour urine oxalate from baseline to after 5 days on low oxalate diet (2 days on participant managed, 3 days on clinical research center prepared diet of 50mg/day) | 6 days
  24-hour urine oxalate will be measured before and after participants follow a low oxalate diet for 5 total days (3 days will be clinical research center prepared food with known measured oxalate content of 50mg/day)
Percent absorption of 13C2-oxalate from pre-load baseline (time 0) to 2, 4-, 6-, and 24-hour time points | 6 days
  Will be measured or calculated at time points 0, 2-hours, 4-hours, 6-hours and 24-hours after sodium 13C2-oxalate and sucralose consumption. We will compare change in urine total urine oxalate and 13C2-oxalate/total oxalate and sucralose each time period for all participants.
Change in urine 13C2-oxalate from pre-load baseline (time 0) to 2, 4-, 6-, and 24-hour time points | 6 days
  Will be measured or calculated at time points 0, 2-hours, 4-hours, 6-hours and 24-hours after sodium 13C2-oxalate and sucralose consumption. We will compare change in urine total urine oxalate and 13C2-oxalate/total oxalate and sucralose each time period for all participants.
Percent absorption total urine oxalate from pre-load baseline (time 0) to 2, 4-, 6-, and 24-hour time points | 6 days
  Will be measured or calculated at time points 0, 2-hours, 4-hours, 6-hours and 24-hours after sodium 13C2-oxalate and sucralose consumption. We will compare change in urine total urine oxalate and 13C2-oxalate/total oxalate and sucralose each time period for all participants.
Percent absorption of sucralose from pre-load baseline (time 0) to 2, 4-, 6-, and 24-hour time points | 6 days
  Will be measured or calculated at time points 0, 2-hours, 4-hours, 6-hours and 24-hours after sodium 13C2-oxalate and sucralose consumption. We will compare change in urine total urine oxalate and 13C2-oxalate/total oxalate and sucralose each time period for all participants.
Change in urine sucralose from pre-load baseline (time 0) to 2, 4-, 6-, and 24-hour time points | 6 days
  Will be measured or calculated at time points 0, 2-hours, 4-hours, 6-hours and 24-hours after sodium 13C2-oxalate and sucralose consumption. We will compare change in urine total urine oxalate and 13C2-oxalate/total oxalate and sucralose each time period for all participants.

SECONDARY OUTCOMES:
Compare change in urine oxalate levels from baseline to post-low oxalate diet between the three groups: lean kidney stone patients, obese kidney stone patients, and post- Roux-en-Y gastric bypass kidney stone patients | 6 days
  1. 24-hour urine oxalate will be measured before and after participants follow a low oxalate diet for 5 total days (3 days will be clinical research center prepared food with known measured oxalate content of 50mg/day).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States